CLINICAL TRIAL: NCT06200363
Title: A Clinical Study of Intravenous MVR-T3011 (T3011) in Combination With Oral Regorafenib in Patients With Advanced Colorectal Cancer
Brief Title: A Clinical Study of T3011 in Combination With Regorafenib in Patients With Advanced Colorectal Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Meng Qiu, Prof., West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MVR-T3011-ES-EC61-CRC
Record Dates: First submitted 2023-10-12; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-12

CONDITIONS: Advanced Colorectal Cancer
MeSH Terms: interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T3011 + Regorafenib (Experimental)
  Interventions: Drug: T3011; Drug: Regorafenib

INTERVENTIONS:
Drug: T3011 — T3011 will be administered intravenously on D1, 4, 8, 11, 15, 18 of each 28-day cycle.
Drug: Regorafenib — Regorafenib will be administered orally once daily for the first 21 days of each 28-day cycle according to NCCN and CSCO guidance.

SUMMARY:
This is a prospective, open, single-arm, investigator-initiated clinical study to evaluate the safety and efficacy of intravenous administration of T3011 at different doses in combination with oral regorafenib in the treatment of advanced colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age ≥ 18 years and ≤ 75 years at the time of informed consent.
2. Histologically or cytologically confirmed advanced unresectable or metastatic colorectal cancer;
3. Anticipated life expectancy ≥3 months
4. At least one measurable lesion per RECIST1.1 criteria, and the lesion has not been treated with radiotherapy before (unless there is definite progression of the lesion after radiotherapy), the longest diameter of the lesion assessed by CT or MRI at baseline is ≥10 mm (the short axis of the lymph node is ≥15 mm); previously received at least second-line or higher standard treatment for advanced colorectal cancer;
5. ECOG performance status 0-2 (including threshold);
6. Weight ≥40kg
7. Hematology:

   * White blood cell (WBC) ≥ 3.0×10^9/L;
   * Neutrophil (ANC) ≥ 1.5×10^9/L;
   * Platelet (PLT) ≥ 75×10^9/L;
   * Hemoglobin (Hb) ≥ 8.0g/dL
8. Hepatic and renal function:

   * Total bilirubin ≤ 1.5 × ULN;
   * Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 2.5 × ULN for patient without liver metastasis, ≤ 5 × ULN for patients with liver metastasis;
   * Serum creatinine ≤ 1.5×ULN, or creatinine clearance ≥ 50 mL/min as determined by the Cockcroft-Gault equation;
9. Coagulation:

   * INR≤1.5 x ULN;
   * APTT≤1.5 x ULN;
10. Women of childbearing potential (WCBP) must have a negative serum pregnancy test at Screening within 14 days of dosing. WCBP, as well as male patients with partners of WCBP, should consent to use at least one medically approved contraceptive method (e.g. surgical sterilization, oral contraceptives, intrauterine devices, abstinence or barrier contraception combined with spermicides) during the study treatment period and for at least 6 months after the last trial drug treatment;
11. Willingness to attend this study, to sign informed consent, to have good compliance, and to cooperate with follow-up visit.

Exclusion Criteria:

1. Pregnant or lactating, or plan to pregnant or give birth during the trial;
2. Persistent or active infection that are not controlled by treatment including but not limited to: active tuberculosis, non-negative HIV antibody, HBsAg positive and HBV DNA ≥LOQ, HCV ab positive and HCV DNA ≥LOQ;
3. Patients with imaging confirmed brain metastasis or brain metastasis history (except patients with stable disease within 3 months before screening and not require systemic glucorticoid therapy according to PI), pia meningeal disease, spinal cord compression;
4. Autoimmune disease or related symptoms, or previously suffered from autoimmune disease;
5. History of splenectomy or organ transplantation;
6. Prior treatment with Oncolytic virus (OV) (including but not be limited to T-VEC), gene therapy, cellular therapy or tumor vaccines;
7. Requires continued concurrent oral or intravenous therapy with any drug against HSV (acyclovir, valaciclovir, penciclovir, famciclovir, ganciclovir, foscarnet, cidofovir). Topical use of drugs against HSV are allowed;
8. Patients plan to receive other anti-tumor therapy (including but not limited to chemotherapy, targeted therapy, immunotherapy, anti-tumor Chinese herbal therapy, etc.) during the study;
9. Patients with a known psychiatric disorder that would interfere with cooperation with the requirements of the trial;
10. History of narcotics (recreational use) and substance abuse (including alcohol) within 1 year prior to signing informed consent;
11. History of allergic reactions attributed to compounds of similar biological composition to HSV-1, IL-12, or anti-PD-1 monoclonal antibody or any excipients for T3011;
12. History or evidence of high risk cardiovascular disease, including but not limited to:

    * Severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, II-III degree atrioventricular block, QT interval corrected using the Fridericia formula (QTcF) ≥ 450 msec (male) or ≥ 470 msec (female);
    * Acute myocardial infarction, unstable angina pectoris, or stroke occurred within 6 months before the first administration of the experimental drug;
    * Coronary angioplasty or stent implantation within 6 months prior to first administration of the experimental drug;
    * Rating of heart function as defined by the New York Heart Association (NYHA) standards>grade II; Cardiac valve abnormalities recorded by echocardiography (≥ grade 2). Note: Subjects with grade 1 cardiac valve abnormalities (such as mild regurgitation/stenosis) were admitted, but subjects with moderate valve thickening were excluded;
    * Left ventricular ejection fraction (LVEF) < the center lower limit. If no lower limit existed, LVEF˂50%;
    * Poor blood pressure control after antihypertensive treatment (i.e. systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg);
13. History of another malignant tumor, except the following:

    * Undergone potentially curative therapy and for ≥5 years prior to the first dose of study treatment and no malignancies with known active disease and low potential recurrence risk;
    * Adequately treated non-melanoma skin cancer or lentigo with no evidence of malignancy;
    * Adequately treated carcinoma in situ without evidence of disease;
14. Received live and attenuated vaccines within 4 weeks prior to initiation of study treatment, or plan to be vaccined during the study;
15. Previous history of immunotherapy induced non-infectious pneumonitis/interstitial lung disease (including but not limited to ≥3 grade irAE) or intolerance to immunotherapy (including but not limited to anti-PD-(L)1 monoclonal Ab), except endocrine-related irAE that can be stably controlled by hormone replacement therapy;
16. Moderate to large amounts of pleural effusion, pericardial effusion, or ascites requiring drug or medical intervention (Patient may be eligible to participate following discussion with investigator and approval from the sponsor);
17. Unexplained >38.5℃ fever (except for tumor induced fever judged by PI) occurs during the screening period, baseline period or on the day of administration, which in the judgment of investigator, would interfere with patient participation in the study or patient's efficacy evaluation;
18. Any condition that PI considered may confuse the trial results, interfere with the patient's participation in the trial, or is not in the participant's best interest to participate in the trial, or a history of treatment or laboratory abnormalities, or other ineligibility for enrollment.

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Adverse event | 28 days after EOT
  To evaluate the safety of intravenous T3011 in combination with oral regorafenib in the treatment of patients with advanced colorectal cancer.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Every 8 weeks until disease progression, consent withdraw, death or end of study, assessed up to 24 months.
  To evaluate the efficacy of intravenous T3011 combined with oral regorafenib in the treatment of patients with advanced colorectal cancer (ORR will be assessed according to RECIST 1.1 & iRECIST)
Disease control rate (DCR) | Every 8 weeks until disease progression, consent withdraw, death or end of study, assessed up to 24 months.
  To evaluate the DCR of intravenous T3011 combined with oral regorafenib in the treatment of patients with advanced colorectal cancer (DCR will be assessed according to RECIST 1.1 & iRECIST)
Progression-free Survival (PFS) | Every 8 weeks until disease progression, consent withdraw, death or end of study, assessed up to 24 months.
  To evaluate the PFS of intravenous T3011 combined with oral regorafenib in the treatment of patients with advanced colorectal cancer (PFS will be assessed according to RECIST 1.1 & iRECIST)
Overall survival (OS) | 24 months
  To evaluate the OS of intravenous T3011 combined with oral regorafenib in the treatment of patients with advanced colorectal cancer
Quality of life questionnaire (QLQ-C30) | Up to 24 months
  The EORTC Core Questionnaire (QLQ-C30) is widely used to measure quality of life in oncology. For self-reported general health and psychological distress, a higher score indicated worse health.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China